CLINICAL TRIAL: NCT01411826
Title: Online Programs to Promote Colon Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kevin Hwang, MD, Assistant Professor - Internal Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSC-MS-11-0305
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Colon Cancer Screening
Keywords: Colon cancer screening
MeSH Terms: interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Information (Active Comparator)
  Interventions: Behavioral: Information Only
- Information + Narratives + Support group (Experimental)
  Interventions: Behavioral: Information + Narratives + Support Group

INTERVENTIONS:
Behavioral: Information + Narratives + Support Group — Information from CDC website Narratives about CRCS written by others Peer social support among study participants
  Arms: Information + Narratives + Support group
Behavioral: Information Only — Information from CDC website on colon cancer screening.
  Arms: Information

SUMMARY:
To evaluate online peer support and colorectal cancer screening behavior among individuals who are not currently meeting colorectal cancer screening guidelines. This is a randomized controlled trial.

DETAILED DESCRIPTION:
Participants in the control group will view standard online information about colon cancer screening. Participants in the intervention group will view the same information and also will be invited to sign on to the online website and interact with peer supporters at their convenience. They will have 6 months to communicate with peer supporters. Peer supporters are encouraged to address comments and concerns of the study participants.

About 300 study participants, majority white, female. Inclusion criteria: age 50-75, not currently meeting colorectal cancer screening guidelines, no previous colorectal cancer.

The study will also include 15 previously identified peer supporters.

Recruitment: Administrators of the SparkPeople.com weight loss community will send study recruitment emails to members at least 50 years of age. Interested individuals will pass an eligibility screening and provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-75
2. Not currently meeting colorectal cancer screening guidelines
3. No previous colorectal cancer.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 months
  Feasibility of recruitment, randomization, intervention delivery, retention, and assessment of colon cancer screening status

SECONDARY OUTCOMES:
Colon cancer screening attitudes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hwang, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Hwang KO, Ottenbacher AJ, Graham AL, Thomas EJ, Street RL Jr, Vernon SW. Online narratives and peer support for colorectal cancer screening: a pilot randomized trial. Am J Prev Med. 2013 Jul;45(1):98-107. doi: 10.1016/j.amepre.2013.02.024. PMID 23790994